CLINICAL TRIAL: NCT00001990
Title: An Open-Label, Uncontrolled Clinical Trial of Oral 566C80 for the Treatment of Patients With Severe PCP Who Are Intolerant and/or Unresponsive to Therapy With Trimethoprim/Sulfamethoxazole and Parenteral Pentamidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 053D; 33384-10
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-04

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Pneumonia, Pneumocystis carinii; Pentamidine; Antifungal Agents; Acquired Immunodeficiency Syndrome; atovaquone
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Atovaquone

INTERVENTIONS:
Drug: Atovaquone

SUMMARY:
To facilitate provision of atovaquone (566C80) to patients who have severe Pneumocystis carinii pneumonia (PCP) and are intolerant and/or unresponsive to trimethoprim / sulfamethoxazole ( TMX / SMX ); to monitor serious adverse events attributable to 566C80.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Clinical diagnosis of acute severe Pneumocystis carinii pneumonia (PCP).
* Dose-limiting intolerance to TMP / SMX and parenteral pentamidine.
* Willingness and ability to give informed consent.

Exclusion Criteria

Co-existing Condition:

Excluded:

* Patients with a history of intolerance to 566C80. Patients with the following prior conditions are excluded: History of serious dose-limiting adverse experience during previous 566C80 therapy, thought to be attributable to the drug.

Required:

* Trimethoprim / sulfamethoxazole (TMP/SMX); pentamidine.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States